CLINICAL TRIAL: NCT07017751
Title: The Effect of Education on Symptom Burden, Medication Adherence, Nutritional Behaviour in Patients With Heart Failure
Brief Title: The Effect of Education on Symptom Burden, Medication Adherence, and Nutritional Behaviour
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Naile ALANKAYA (Other)
Responsible Party: Sponsor-Investigator, Naile ALANKAYA, Assoc. Prof., Çanakkale Onsekiz Mart University
Organization: Çanakkale Onsekiz Mart University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMU-SBF-NA-02
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Heart Diseases; Heart Failure
Keywords: Symptom Burden; Medication Adherence; Nutritional Behaviour; heart failure
MeSH Terms: conditions — Heart Diseases; Heart Failure; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervetion group (Experimental): The intervention group will consist of 30 people. The intervention group will receive 45 minutes online education structured according to Pender's Health Promotion Model on symptom burden, medication adherence, and nutritional behaviour in patients with heart failure. Two weeks, one month, and two months after the initial education, participants will be contacted to obtain feedback on their post-education dietary behaviours, medication compliance, and symptoms.
  Interventions: Other: Heart failure medication
- Control group (No Intervention): The control group will consist of 30 people. All patients will be asked to complete the Heart Failure Symptom Status Scale, Medication Adherence and Prescription Writing Scale. Patients in the control group will not receive any training. The same forms will be filled out for the final test 3 months later. Patients who wish to will be given the training provided in the experimental group.

INTERVENTIONS:
Other: Heart failure medication — intervention group will receive 45 minutes online education structured according to Pender's Health Promotion Model on symptom burden, medication adherence, and nutritional behaviour in patients with heart failure. Two weeks, one month, and two months after the initial education, participants will be contacted to obtain feedback on their post-education dietary behaviours, medication compliance, and symptoms.
  Other Names: Heart Failure training
  Arms: Intervetion group

SUMMARY:
This study aims to determine the effect of online education structured according to Pender's Health Promotion Model on symptom burden, medication adherence, and nutritional behaviour in patients with heart failure. The sample size was calculated using the 'G. Power-3.1.9.2' programme at a 95% confidence level prior to data collection. Accordingly, the minimum sample size required for the independent sample t-test for the study was determined to be 44 (22 for each group) based on an alpha value of 0.05, an effect size of 1.128, and a theoretical power of 95%. Taking data losses into account, a total of 60 patients (30 for each group) were planned to be included in the sample. Data will be collected using the Heart Failure Symptom Status Scale, Medication Adherence and Prescription Printing Scale (İURYÖ-7), Heart Failure Nutrition Behaviour Scale. 1: Prior to providing education to patients, they will be informed about the purpose of the study, the data collection method, and the topics to be covered in the education. Patients who agree to participate in the study will be asked to sign an informed consent form. All patients in the experimental and control groups will be asked to complete the Heart Failure Nutrition Behaviour Scale (HFNBS), Heart Failure Symptom Status Scale (HFSSS), and Medication Adherence and Prescription Writing Scale (MAPWS-79) before receiving education.

2: The contact information of all patients in the experimental group will be collected. Training will be provided online at a time and date convenient for the patients.

3: Patients in the control group will receive a digital training booklet prepared by the researcher at the contact address they provide.

4: Participants will be contacted 2 weeks, 1 month, and 2 months after the initial education session to obtain feedback on post-education dietary behaviours, medication adherence, and symptoms.

5: Four to six weeks after the training is completed, the 'Nutritional Behaviour Scale in Heart Failure,' 'Heart Failure Symptom Status Scale,' and 'Medication Adherence and Prescription Writing Scale (İURYÖ-7)' will be completed online again. The same forms will also be completed online by patients in the control group 4-6 weeks later.

DETAILED DESCRIPTION:
Heart failure (HF) is emerging as a major public health problem worldwide. As a chronic and progressive disease, HF reduces individuals' quality of life and places a significant burden on healthcare systems. Heart failure is becoming more prevalent, particularly with an ageing population, and is increasing morbidity and mortality rates. In this context, effective management of HF and improvement of patient outcomes require a multidisciplinary approach.

Adherence to appropriate treatment and adoption of healthy lifestyle behaviours are critical in slowing disease progression and reducing the risk of complications in patients with HF. However, the literature reports that HF patients have low treatment adherence rates and experience difficulties in implementing lifestyle changes. In particular, poor medication adherence and unhealthy eating habits increase readmission rates and negatively impact patients' overall health.

Factors contributing to low medication adherence and unhealthy dietary behaviours in CF patients include symptom burden, lack of knowledge about the disease, low self-efficacy, perceived barriers, and lack of social support. This situation highlights not only the inadequacy of biomedical treatment approaches but also the need for education and support programmes that target individuals' behavioural determinants. Pender's Health Promotion Model provides an effective framework in this context. The model focuses on individual characteristics, behavioural determinants, and outcome behaviours that influence individuals' adoption of health behaviours. Identifying factors such as self-efficacy, perceived benefits, and barriers is an important starting point for behavioural change. In recent years, online support lines and digital health technologies have emerged as a promising approach in chronic disease management. Online education and support programmes for HFpatients have the potential to increase treatment adherence, improve symptom management, and encourage healthy lifestyle changes. Online support can enhance individuals' self-efficacy and reduce social support deficits, particularly among HF patients, by facilitating access to information. However, there are limited studies in the literature regarding the effectiveness of such programmes, and most existing studies are not grounded in a theoretical framework such as Pender's model.

A better understanding of the factors influencing medication adherence and dietary behaviour in HF patients and an evaluation of the role of online support lines in this context could provide significant benefits at both the individual and societal levels. An approach based on Pender's Health Behaviour Change Model can address not only individuals' behavioural changes but also the underlying psychosocial factors driving these changes. In this regard, studies evaluating the effectiveness of online support lines for HF patients are expected to make significant contributions to both scientific knowledge and healthcare practices.

This study aims to determine the effect of online education structured according to Pender's Health Promotion Model on symptom burden, medication adherence, and nutritional behaviour in patients with heart failure.

This study was designed as a randomised controlled trial to determine the effect of online education structured according to Pender's Health Development Model on symptom burden, medication adherence, and dietary behaviour in patients with heart failure.

The sample size required for randomisation into groups was calculated prior to data collection using the 'G. Power-3.1.9.2' programme at a 95% confidence level. Accordingly, the minimum sample size required for the independent sample t-test for the study was determined to be 44 (22 per group) using an alpha value of 0.05, an effect size of 1.128, and a theoretical power of 95%. Considering data losses, a total of 60 patients (30 per group) were planned to be included in the sample.Before educating patients, information will be provided about the purpose of the study, the data collection method, and the topics to be covered in the education. Patients who agree to participate in the study will be asked to sign an informed consent form. Data collection will take place in two stages.

1. Stage: All patients (experimental and control) will be asked to complete the Heart Failure Symptom Status Scale, Medication Adherence and Prescription Writing Scale. Individual education will be conducted online for patients in the experimental group at a suitable time and date. The education will be conducted via applications such as WhatsApp or Google Meet. In addition, a digital education booklet and a video of the education will be sent to the patients' contact addresses. Patients in the control group will only be given the digital education booklet.
2. Two weeks, one month, and two months after the initial education, participants will be contacted to obtain feedback on their post-education dietary behaviours, medication compliance, and symptoms.

Four to six weeks after the training is completed, the experimental group will again complete the 'Nutritional Behaviour Scale in Heart Failure,' 'Heart Failure Symptom Status Scale,' and 'Medication Adherence and Prescription Writing Scale (İURYÖ-7)' online. The same forms will also be completed online by patients in the control group 4-6 weeks later. Additionally, the video prepared for the experimental group will be shared with the control group.

Data Collection Tools Data will be collected using the Heart Failure Symptom Status Scale, Medication Adherence and Prescription Printing Scale (İURYÖ-7), and Heart Failure Nutrition Behaviour Scale.

The universe of the study consisted of patients diagnosed with heart failure who applied to Dr. Burhan Nalbantoğlu Hospital.

Inclusion Criteria:

* Diagnosed with heart failure,
* 18 years of age or older,
* Access to the internet and the technical infrastructure to participate in online training,
* Voluntarily agreeing to participate in the study.

Exclusion Criteria:

* Having severe cognitive or psychological disorders,
* Having difficulty communicating,
* Being in the process of heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Diagnosed with heart failure.
* Not having cognitive dysfunction.
* Access to the internet and the technical infrastructure to participate in online training.

Exclusion Criteria:

* Having severe cognitive or psychological disorders,
* Having difficulty communicating,
* Being in the process of heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Heart Failure Symptom Status Scale | Baseline and after 6 months
  The scale addresses seven primary symptoms: dyspnoea, dyspnoea when lying supine, fatigue, chest pain, oedema, sleep problems, dizziness, and loss of balance.The total score that can be obtained from the scale ranges from 0 to 84. An increase in the score indicates a greater symptom burden.
Medication Adherence and Prescription Writing Scale | Baseline and after 6 months
  The scale can also be used to determine medication adherence in individuals with low literacy levels. The scale consists of two subscales: the medication adherence subscale ranges from 4 to 16 points, and the prescription subscale ranges from 3 to 12 points. Item 7 is reverse-coded in the scale.The scale consists of 7 items, with the lowest possible score being 7 and the highest possible score being 28. As the score obtained from the scale decreases, medication adherence increases.
Heart Failure Nutrition Behaviour Scale | Baseline and after 6 months
  The HFNBS consists of four subscales: healthy habits, salt restriction, sugar restriction, and prevention of retention, and comprises a total of 19 items. . A high total score on the scale indicates that individuals have adopted a diet consistent with the recommended dietary guidelines for heart failure; a low score indicates that individuals are not following these recommendations. The interpretation of the scores is as follows:
  * 19 ≤ score <46: Patients are not following the guidelines and expert recommendations.
  * 46 ≤ score <51: Patients are following the guidelines and expert recommendations to some extent.
  * 51 ≤ score <55: Patients are following the guidelines and expert recommendations to a moderate extent.
  * 55 ≤ score ≤76: Patients are following the guidelines and expert recommendations to a high extent.

CONTACTS AND LOCATIONS:
Overall Officials: NAİLE ALANKAYA, Assoc. Prof, Study Director — Çanakkale Onsekiz Mart University, Faculty of Health Sciences
Locations (1):
- Çanakkale Onsekiz Mart University, Faculty of Health Sciences, Merkez, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No